CLINICAL TRIAL: NCT05230654
Title: Efficacy and Safety of Fosaprepitant in Preventing Chemotherapy-induced Vomiting in Children Treated With Medium and High Emetic Chemotherapeutic Drugs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: fosaprepitant
Record Dates: First submitted 2022-01-28; First posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Chemotherapy Induced Nausea and Vomiting Pediatric Cancer Patients
Keywords: Fosaprepitant; Chemotherapy-induced nausea and vomiting; Pediatric patients; Emetogenic chemotherapy
MeSH Terms: conditions — Vomiting | interventions — fosaprepitant

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fosaprepitant (Experimental): Patients received intravenous Ganisetron plus dexamethasone followed by fosaprepitant infusion
  Interventions: Drug: Fosaprepitant
- Placebo (Placebo Comparator): Patients received intravenous Ganisetron plus dexamethasone followed by normal saline
  Interventions: Drug: Placebo(normal saline)

INTERVENTIONS:
Drug: Fosaprepitant — Fosaprepitant: 4 mg/kg IV Granisetron+dexamethasone: granisetron:40mcg/kg, IV ; dexamethasone : S<0.6m2, 2 mg/dose, q12h IV/PO; S>0.6m2, 4 mg/dose, q12h , IV/PO. When used with fosaprepitant, dexamethasone dose was halved.
  Arms: fosaprepitant
Drug: Placebo(normal saline) — Placebo(normal saline): 4 ml/kg IV Granisetron+dexamethasone: granisetron:40mcg/kg, IV ; dexamethasone : S<0.6m2, 2 mg/dose, q12h IV/PO; S>0.6m2, 4 mg/dose, q12h , IV/PO.
  Arms: Placebo

SUMMARY:
This study was a prospective, randomized, double-blind, parallel controlled clinical trial. The children who met the inclusion criteria and were treated with medium and high emetic chemotherapy drugs were randomly included in the experimental group (forsapitan group) and the control group (placebo group) in the ratio of 1 ∶ 1. The children in the experimental group were infused with fosapitan, dexamethasone and granisetron before chemotherapy, and then continued to be infused with granisetron and dexamethasone until 48 hours after the end of chemotherapy. The antiemetic regimen of children in the control group was placebo instead of fosapitan, and the others were the same as those in the experimental group. In this study, CNNC antiemetic scale and pediatric scale proposed by Dupuis were used to evaluate the vomiting data. The primary end point was the proportion of children who achieved complete remission (CR) in the delayed period (within 24-120 hours after the start of chemotherapy); The secondary end points were the CR rate in the acute phase (within 24 hours after the first chemotherapy administration) and the overall phase. The antiemetic efficacy and adverse reactions of the two groups were observed and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* children aged 2-12 years at the time of study entry with documented cancer scheduled to receive MEC or HEC (more than 30% emetogenic potential) with Karnofsky score of 60 or more (for patients aged greater than 10 years) or Lansky play performance score of 60 or more (for patients aged 10 years or less) predicted life expectancy of at least 3 months; and written informed consent provided by parent or guardian

Exclusion Criteria:

* vomiting 24 hours before treatment day 1 known history of QT prolongation or allergic reaction to any of the study drugs symptomatic primary or metastatic CNS malignancy causing nausea or vomiting patients who received radiation therapy to the abdomen or pelvis in the week before treatment; active infection or any uncontrolled concurrent illness except for malignancy abnormal laboratory values at screening (peripheral absolute neutrophil count <1000 cells per μL, platelet count <100 000 cells per μL; alanine amino transferase or aspartate aminotransferase >5 times of the upper limit of normal for age, bilirubin or serum creatinine >1.5 times of the upper limit of normal for age) initiation of systemic corticosteroids within 72 hours before study drug administration or as part of the chemotherapy regimen; benzodiazepines or opioids initiated within 48 hours before treatment, except for single doses of triazolam, temazepam, or midazolam use of antiemetics within 48 hours of treatment use of CYP3A4 substrates or inhibitors within 7 days or CYP3A4 inducers within 30 days of treatment

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Complete remission rates in the acute phases | up to 6 months
  The primary end point was complete remission rates in the acute phase. Complete Remission was defined as no vomiting, no retching, and no use of rescue medecation

SECONDARY OUTCOMES:
Complete Remission rates in the delayed and overall phases | up to 6 months
  Complete Remission rates in the delayed and overall phases
Adverse events reported in study patients | up to 6 months
  All of the adverse reaction of aprepitant and fosaprepitant during the study

CONTACTS AND LOCATIONS:
Overall Officials: Yijin Gao, Study Director — Shanghai Children's Medical Center
Locations (1):
- Shanghai Children's Medical Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flank J, Robinson PD, Holdsworth M, Phillips R, Portwine C, Gibson P, Maan C, Stefin N, Sung L, Dupuis LL. Guideline for the Treatment of Breakthrough and the Prevention of Refractory Chemotherapy-Induced Nausea and Vomiting in Children With Cancer. Pediatr Blood Cancer. 2016 Jul;63(7):1144-51. doi: 10.1002/pbc.25955. Epub 2016 Mar 9. PMID 26960036
- [Background] Weinstein C, Jordan K, Green SA, Camacho E, Khanani S, Beckford-Brathwaite E, Vallejos W, Liang LW, Noga SJ, Rapoport BL. Single-dose fosaprepitant for the prevention of chemotherapy-induced nausea and vomiting associated with moderately emetogenic chemotherapy: results of a randomized, double-blind phase III trial. Ann Oncol. 2016 Jan;27(1):172-8. doi: 10.1093/annonc/mdv482. Epub 2015 Oct 8. PMID 26449391
- [Background] Radhakrishnan V, Joshi A, Ramamoorthy J, Rajaraman S, Ganesan P, Ganesan TS, Dhanushkodi M, Sagar TG. Intravenous fosaprepitant for the prevention of chemotherapy-induced vomiting in children: A double-blind, placebo-controlled, phase III randomized trial. Pediatr Blood Cancer. 2019 Mar;66(3):e27551. doi: 10.1002/pbc.27551. Epub 2018 Nov 13. PMID 30426714
- [Background] Mora J, Valero M, DiCristina C, Jin M, Chain A, Bickham K. Pharmacokinetics/pharmacodynamics, safety, and tolerability of fosaprepitant for the prevention of chemotherapy-induced nausea and vomiting in pediatric cancer patients. Pediatr Blood Cancer. 2019 Jun;66(6):e27690. doi: 10.1002/pbc.27690. Epub 2019 Mar 21. PMID 30900392
- [Background] Dupuis LL, Boodhan S, Holdsworth M, Robinson PD, Hain R, Portwine C, O'Shaughnessy E, Sung L; Pediatric Oncology Group of Ontario. Guideline for the prevention of acute nausea and vomiting due to antineoplastic medication in pediatric cancer patients. Pediatr Blood Cancer. 2013 Jul;60(7):1073-82. doi: 10.1002/pbc.24508. Epub 2013 Mar 19. PMID 23512831